CLINICAL TRIAL: NCT04539860
Title: Comparison of Blood Pressure Measurements Between Transdermal Optical Imaging and Standard of Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Nuralogix Corporation (Industry); The Affiliated Hospital of Hangzhou Normal University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Kang Lee, Professor, University of Toronto
Other Study IDs: 32755
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Blood pressure measurements by standard assessment methods and Transdermal Optical Imaging
  Interventions: Device: Transdermal Optical Imaging
- Patients: Blood pressure measurements by standard assessment methods and Transdermal Optical Imaging
  Interventions: Device: Transdermal Optical Imaging

INTERVENTIONS:
Device: Transdermal Optical Imaging — Blood pressure measurements completed by standard assessment methods and Transdermal Optical Imaging

SUMMARY:
Participants (patients and volunteers) will be recruited to have their blood pressure measured by standard blood pressure assessment methods while having their face video recorded. The data collected will help improve the blood pressure measurement accuracy of Transdermal Optical Imaging, which relies on machine learning to extract physiological information from videos recorded.

DETAILED DESCRIPTION:
There are many ways to measure blood pressure (monitors, mercury sphygmomanometer, aneroid devices), with most relying on a cuff-inflation. Transdermal Optical Imaging measures blood pressure using a video captured by any conventional camera (e.g., those on a phone, tablet, laptop) and advanced machine learning algorithms.

The current study aims to improve the accuracy of Transdermal Optical Imaging algorithms for measuring blood pressure. The investigators will recruit participants (patients with medical problems and healthy volunteers) to have their blood pressure measured in various ways (e.g.,by registered nurses with sphygmomanometer and stethoscope, continuous blood pressure monitor, etc.). Further, participants will have their faces video-recorded intermittently between standard measurements or at the same time as standard measures.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent to participate (including by parent or legal guardian if under 16 years old).

Exclusion Criteria:

* No exclusion criteria

Ages: 13 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Only individuals, of any sex, over the age of 13 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Results | Single visit; up to one day
  Comparison of Transdermal Optical Imaging data and Standard assessment data

CONTACTS AND LOCATIONS:
Overall Officials: Kang Lee, PhD, Principal Investigator — University of Toronto
Locations (3):
- University of Toronto, Toronto, Ontario, Canada
- China (2):
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers outside the team of researchers involved in the current study. Findings of the study based on group results will be shared in publications.